CLINICAL TRIAL: NCT02248688
Title: Gastric Artery Embolization Trial for Lessening Appetite Nonsurgically (GET LEAN)
Brief Title: Gastric Artery Embolization Trial for Lessening Appetite Nonsurgically
Acronym: GETLEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dayton Interventional Radiology (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Q131650
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Arterial Embolization; Other Surgical Procedures; Obesity
Keywords: Bariatric Embolization; Gastric Artery Emboliziation; Left Gastric Artery Embolization; Morbid Obesity; Obesity; Weight Loss; Ghrelin; Embolization
MeSH Terms: conditions — Obesity; Obesity, Morbid; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Embolic Agent - BeadBlock (Other): Left Gastric Artery Embolization - Embolic Agent - BeadBlock 300 - 500 Micron will be used as the embolic agent to embolize left gastric artery.
  Interventions: Device: BeadBlock 300 - 500 Micron; Procedure: Left Gastric Artery Embolization

INTERVENTIONS:
Device: BeadBlock 300 - 500 Micron — Beadblock will be used intraarterially to occlude the left gastric artery and its branches. The left gastric artery supplies the fundus of the stomach, where it is known that the hormone Ghrelin (one of the hormones responsible for appetite) is produced.
  Other Names: GET LEAN
Procedure: Left Gastric Artery Embolization

SUMMARY:
The purpose of this pilot study is to achieve the collection of safety and efficacy data in patients undergoing left gastric artery embolization for morbid obesity in the United States. As secondary goal, the pilot study seeks to obtain quality of life data. This pilot study is not designed to achieve new indications for this device.

DETAILED DESCRIPTION:
Beadblock will be used intraarterially to occlude in this case the left gastric artery and its branches. The left gastric artery supplies the fundus of the stomach, where it is known that the hormone ghrelin (one of the hormones responsible for appetite) is produced. Ghrelin is a 28 amino acid hunger stimulating peptide and hormone that is produced mainly by P/D1 cells lining the fundus of the stomach and epsilon cells of the pancreas. Ghrelin has emerged as the first identified circulating hunger hormone. Ghrelin is also the only known circulating orexigen, or appetite enhancing hormone.

Left gastric artery embolization may be a minimally invasive alternative to the current surgical treatment of gastric bypass or reduction surgery. These treatments have known serious complications including anastomotic leaks, bowel obstruction, paralytic ileus, deep vein thrombosis, pulmonary embolism, gastrointestinal bleeding, dumping syndrome, and anesthesia risks resulting in morbidity and mortality.

Literature review for gastric artery embolization

Transarterial embolization is a common interventional procedure used to treat a variety of medical conditions. In the image-guided procedure, an embolic, or obstructive, agent is inserted through a catheter and placed inside an artery to prevent blood flow in an artery or to a specific area of the body. Types of embolic agents include beads, coils, gel foam,as well as other materials and devices.

Gastric artery embolization has been used since the 1970's to treat life threatening gastric hemorrhage. This is commonly accepted as standard of care and has been life saving for thousands of patients. It is even deemed to be effective enough to be used empirically in the setting of angiographically negative life threatening hemorrhage (as a reflection of its safety margin).

Recent animal studies over the past several years in porcine and canine models have shown that gastric artery embolization results in the suppression of ghrelin levels and weight loss.

Arepally, et al. (2008) first described the technique of gastric artery embolization to reduce weight gain. In a controlled study, he used sodium morrhuate within a porcine model with resultant lower ghrelin levels and significantly blunted weight gain (in otherwise rapidly growing young swine).

Paxton, et al. (SIR abstract in 2012, later published in 2013 and 2014) described the technique of 40 micron microsphere particle embolization in a similar porcine model that also resulted in lowered ghrelin levels and reduced weight gain. Also noted there was no duodenal upregulation for ghrelin.

Bawudun et al. (2012) described a technique of left gastric embolization using mixture of bleomycin and lipiodol versus polyvinyl alcohol 500-700 micron particles to create weight loss in a canine model without gastric ulceration. In addition, he demonstrated significant reduction in subcutaneous fat and plasma ghrelin.

Kipshidze, et al. (2013) performed the first in man study reported at the annual meeting of the American College of Cardiology that showed an average of 45lbs of weight loss in 6 months and reduced ghrelin levels in 5 patients with no complications (with endoscopic follow-up) in this small series using BeadBlock 300-500 micron particles. According to personal correspondence with the author of this study the weight loss is sustained for at least 1 year with no complications in these 5 patients. He also noted that an additional 7 patients have been treated without complications.

A recent retrospective case control study presented at the 2013 Radiological Society of North American annual meeting found that there was an average of 7.9% decrease in body weight (at 3 months) in 15 patients who underwent left gastric artery embolization for life threatening hemorrhage compared to 1.2% (P=0.001) for age matched controls (who underwent embolization other than the left gastric artery for upper gastrointestinal bleeding).

ELIGIBILITY:
Inclusion Criteria:

Morbid obesity with a BMI ≥ 40 Age ≥ 22years Ability to lay supine on an angiographic table <400lbs due to table weight limits Appropriate anesthesia risk as determined by certified anesthesia provider evaluation preprocedure.

Willing, able and mentally competent to provide written informed consent (to ensure that all study subjects demonstrate an understanding of the risks of the procedure and also participate in the informed consent).

Subjects who have failed previous attempts at weight loss through diet, exercise, and behavior modification (as it is recommended that conservative options, such as supervised low calorie diets combined with behavior therapy and exercise, should be attempted prior to enrolling in this study).

Exclusion Criteria:

Less than 22 years of age Major surgery within the past eight weeks Previous gastric, pancreatic, hepatic and splenic surgery Previous radiation therapy to the left or right upper quadrant Previous gastric, hepatic, or splenic embolization Any history of portal venous hypertension Serum creatinine > 1.8 mg/dL History of kidney problems Pregnant or intend to become pregnant within one year History of severe bleeding disorder (platelet count less than 40,000) Allergy to materials in the embolic agents (acrylamido polyvinyl alcohol macromer) Enrolled in another study Any patient who has a history of allergic reaction to iodinated contrast Abnormal baseline gastric emptying study Patients taking anti-coagulants or antiplatelet drugs Patients currently taking or requiring chronic use of NSAID or steroid medications Patients with any chronic upper gastrointestinal complaints such as pain, nausea or vomiting Patients with any history of peptic ulcer disease Patients with any indication of gastrointestinal bleeding as documented by positive stool guaiac and complete blood count with abnormalities.

Patients with any contraindications for monitored anesthesia care or general surgery Patients with secondary causes of obesity such as Cushing's disease and hypothyroidism Patients with active substance abuse or alcoholism Patients with defined noncompliance with previous medical care Patients with certain psychiatric disorders such as schizophrenia, borderline personality disorder, and uncontrolled depression, and mental/cognitive impairment that limits the individual's ability to understand the proposed therapy.

Subjects with mesenteric atherosclerotic disease or abdominal angina should be excluded due to safety concerns.

Patients with hiatal hernia Patients with known aortic disease, such as dissection or aneurysm Patients with comorbidity such as cancer, peripheral arterial disease or other cardiovascular disease Patients with any abnormality on their baseline EGD Patients with a CT Angiogram demonstrate an anatomical variant in left gastric artery anatomy

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-09; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mubin I Syed, MD, Principal Investigator — Dayton Interventional Radiology; Azim Shaikh, MD, MBA, Study Director — Dayton Interventional Radiology; Sumeet Patel, Study Director — Dayton Interventional Radiology; Feras J Deek, BS, BA, Study Director — Dayton Interventional Radiology
Locations (1):
- Dayton Interventional Radiology, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest left gastric artery embolization for the treatment of morbid obesity. Data shared will be coded, with no PHI included. Approval of the request and is a prerequisite to the sharing of data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP).

REFERENCES:
- [Background] Rosch J, Dotter CT, Brown MJ. Selective arterial embolization. A new method for control of acute gastrointestinal bleeding. Radiology. 1972 Feb;102(2):303-6. doi: 10.1148/102.2.303. No abstract available. PMID 4536688
- [Background] Bookstein JJ, Chlosta EM, Foley D, Walter JF. Transcatheter hemostasis of gastrointestinal bleeding using modified autogenous clot. Radiology. 1974 Nov;113(2):277-85. doi: 10.1148/113.2.277. No abstract available. PMID 4547597
- [Background] Morris DC, Nichols DM, Connell DG, Burhenne HJ. Embolization of the left gastric artery in the absence of angiographic extravasation. Cardiovasc Intervent Radiol. 1986;9(4):195-8. doi: 10.1007/BF02577940. PMID 3094950
- [Background] Arepally A, Barnett BP, Patel TH, Howland V, Boston RC, Kraitchman DL, Malayeri AA. Catheter-directed gastric artery chemical embolization suppresses systemic ghrelin levels in porcine model. Radiology. 2008 Oct;249(1):127-33. doi: 10.1148/radiol.2491071232. PMID 18796671
- [Background] Paxton BE, Alley CL, Crow JH, Burchette J, Weiss CR, Kraitchman DL, Arepally A, Kim CY. Histopathologic and immunohistochemical sequelae of bariatric embolization in a porcine model. J Vasc Interv Radiol. 2014 Mar;25(3):455-61. doi: 10.1016/j.jvir.2013.09.016. Epub 2014 Jan 21. PMID 24462005
- [Background] Paxton BE, Kim CY, Alley CL, Crow JH, Balmadrid B, Keith CG, Kankotia RJ, Stinnett S, Arepally A. Bariatric embolization for suppression of the hunger hormone ghrelin in a porcine model. Radiology. 2013 Feb;266(2):471-9. doi: 10.1148/radiol.12120242. Epub 2012 Nov 30. PMID 23204538
- [Background] Bawudun D, Xing Y, Liu WY, Huang YJ, Ren WX, Ma M, Xu XD, Teng GJ. Ghrelin suppression and fat loss after left gastric artery embolization in canine model. Cardiovasc Intervent Radiol. 2012 Dec;35(6):1460-6. doi: 10.1007/s00270-012-0362-8. Epub 2012 Feb 25. PMID 22367009
- [Background] Brown KT, Friedman WN, Marks RA, Saddekni S. Gastric and hepatic infarction following embolization of the left gastric artery: case report. Radiology. 1989 Sep;172(3):731-2. doi: 10.1148/radiology.172.3.2788892.
- [Background] Castaneda-Zuniga WR, Jauregui H, Rysavy J, Amplatz K. Selective transcatheter embolization of the upper gastrointestinal tract: an experimental study. Radiology. 1978 Apr;127(1):81-3. doi: 10.1148/127.1.81. PMID 305577
- [Background] Bradley EL 3rd, Goldman ML. Gastric infarction after therapeutic embolization. Surgery. 1976 Apr;79(4):421-4. PMID 1083078
- [Background] Prochaska JM, Flye MW, Johnsrude IS. Left gastric artery embolization for control of gastric bleeding: a complication. Radiology. 1973 Jun;107(3):521-2. doi: 10.1148/107.3.521. No abstract available. PMID 4702528
- [Background] Robbins SM, Tuten TU, Clements JL, Fekete P. Angiographic diagnosis of gastric volvulus with report of a complication following left gastric artery embolization. Gastrointest Radiol. 1988;13(2):112-4. doi: 10.1007/BF01889038. PMID 3258835
- [Background] Miller DL, Balter S, Cole PE, Lu HT, Schueler BA, Geisinger M, Berenstein A, Albert R, Georgia JD, Noonan PT, Cardella JF, St George J, Russell EJ, Malisch TW, Vogelzang RL, Miller GL 3rd, Anderson J; RAD-IR study. Radiation doses in interventional radiology procedures: the RAD-IR study: part I: overall measures of dose. J Vasc Interv Radiol. 2003 Jun;14(6):711-27. doi: 10.1097/01.rvi.0000079980.80153.4b. PMID 12817038
- [Background] Syed MI, Morar K, Shaikh A, Craig P, Khan O, Patel S, Khabiri H. Gastric Artery Embolization Trial for the Lessening of Appetite Nonsurgically (GET LEAN): Six-Month Preliminary Data. J Vasc Interv Radiol. 2016 Oct;27(10):1502-8. doi: 10.1016/j.jvir.2016.07.010. Epub 2016 Aug 24. PMID 27567998

RESULTS

PARTICIPANT FLOW:
Groups:
- BeadBlock 300 - 500 Micron Will be Used as the Embolic Agent to Embolize Left Gastric Artery.: Beadblock will be used intraarterially to occlude the left gastric artery and its branches. The left gastric artery supplies the fundus of the stomach, where it is known that the hormone Ghrelin (one of the hormones responsible for appetite) is produced.
Period: Overall Study
Arm/Group | BeadBlock 300 - 500 Micron Will be Used as the Embolic Agent to Embolize Left Gastric Artery.
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Embolic Agent - BeadBlock: Left Gastric Artery Embolization - Embolic Agent - BeadBlock 300 - 500 Micron will be used as the embolic agent to embolize left gastric artery.
  BeadBlock 300 - 500 Micron: Beadblock will be used intraarterially to occlude the left gastric artery and its branches. The left gastric artery supplies the fundus of the stomach, where it is known that the hormone Ghrelin (one of the hormones responsible for appetite) is produced.
  Left Gastric Artery Embolization
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Weight [Mean (Full Range); unit: Pounds] | 242.2 [184 to 275]
BMI [Mean (Full Range); unit: kg/m^2] | 42.42 [40 to 45]
Cholecystokinin [Mean (Full Range); unit: pg/mL] | 55.8 [10 to 101]
Ghrelin [Mean (Full Range); unit: pg/mL] | 794 [391 to 1524]
Leptin [Mean (Full Range); unit: ng/mL] | 30.0 [17.3 to 46.3]
Hemoglobin-A1c (HgA1c) [Number; unit: Percentage of HgA1c] — Applicable to sole diabetic participant. Population: Measure taken for diabetic participant.
  Percentage of HgA1c
    number analyzed (Participants) | 1
    (all) | 7.4
Urine Pregnancy Test (only if female of child-bearing potential) [Number; unit: Number of Participants] — Population: Measure only taken for female participants. A participant who is pregnant (i.e., has a positive urine pregnancy test) will be scored as a "1".
  A participant who is not pregnant (i.e., has a negative urine pregnancy test) will be scored as a "0".
  Number of Participants
    number analyzed (Participants) | 4
    (all) | 0
Complete blood count (CBC) [Count of Participants; unit: Participants] — CBC categorized as normal or abnormal. Normal, defined as results in the following ranges White Blood Cell Count: 3.8-10.8 k/mm^3 Red Blood Cell Count: 3.9-5.2 M/mm^3 Hemoglobin: 12-15.6 g/dL Hematocrits: 35-46% Mean Corpuscular Volumes: 80-100.0 fL Mean Corpuscular Hemoglobin (MCH): 27-33 pg MCH Concentration: 32-36 g/dL Red Cell Distribution Widths: 9-15% Platelet Counts: 130-400 k/mm^3
  Abnormal defined as any of results lying outside the normal ranges described above
  Participants
    Normal | 5
    Abnormal | 0
Blood Urea Nitrogen (BUN)/Creatinine [Count of Participants; unit: Participants] — Categorized as normal or abnormal. Normal defines as a BUN within the range of 3-29 mg/dL and Creatinine 0.5-1.2 mg/dL.
  Abnormal defines as results outside the normal ranges described above.
  Participants
    Normal | 5
    Abnormal | 0
Prothrombin Time/Partial Thromboplastin Time (PT/PTT) [Count of Participants; unit: Participants] — Categorized either as normal or abnormal. Normal defined as an Activated PTT result within the range of 20.0-30.0 seconds and a Prothrombin Time within the range of 9-12.5 seconds.
  Abnormal defines as results outside the normal ranges described above.
  Participants
    Normal | 5
    Abnormal | 0
Computed Tomography (CT) Angiogram [Count of Participants; unit: Participants] — Categorized as normal or abnormal. Normal defined as 1) the left gastric artery (LGA) did not arise from the gastrohepatic trunk and 2) the LGA did not arise directly from the aorta
  Abnormal defined as LGA that did arise from the gastrohepatic trunk or directly from the aorta
  Variant vascular anatomy of the left gastrohepatic trunk was noted in the sole participant with an "abnormal" CT-angiogram. The SureFire anti-flux catheter with embolic protection device was used to avoid possible migration of the bead block to non-targeted areas of intervention.
  Participants
    Normal | 4
    Abnormal | 1
Upper Endoscopy [Count of Participants; unit: Participants] — Categorized as normal or abnormal. Normal defined as presentation normal color and without bleeding, growths, ulcers, or inflammation Abnormal defined as results that are not congruent with the normal results presented above.
  Participants
    Normal | 5
    Abnormal | 0
Stool Guaiac [Count of Participants; unit: Participants] — Categorized as normal or abnormal. Normal defined as a negative hemoccult test Abnormal defined as a postive hemoccult test.
  Participants
    Normal | 5
    Abnormal | 0
Nuclear Medicine: Gastric Emptying Study [Count of Participants; unit: Participants] — Categorized as normal or abnormal. Normal defined as 50% or greater gastric emptying within 60-90 minutes. Abnormal defined as results lying outside the range described above.
  Participants
    Normal | 5
    Abnormal | 0
Short Form (SF)-36v2 Questionnaire, Physical Component Summary (PCS) [Mean (Full Range); unit: Scores on a Scale] — The mean of participant's SF-36 Version 2 PCS, ranging from 0-100; higher scores indicate better health status. The SF-36v2 contains 8 sections total which are each calculated into individual scale scores. A z-score is then determined for each scale score by subtracting the mean scale score of a sample of the national general population from the scale score of the individual participant being analyzed. Each of the 8 z-scores are then multiplied by the PCS scoring coefficient, added together, multiplied by 10 and added to 50.
  Scores on a Scale | 49.8 [36 to 84.5]
Short Form (SF)-36 Version 2 Questionnaire Mental Component Summary (MCS) [Mean (Full Range); unit: Scores on a Scale] — The mean of participant's Short Form-36 Version 2 MCS, ranging from 0-100; higher scores indicate better health status. The SF-36v2 contains 8 sections total which are each calculated into individual scale scores. A z-score is then determined for each scale score by subtracting the mean scale score of a sample of the national general population from the scale score of the individual participant being analyzed. Each of the 8 z-scores are then multiplied by the MCS scoring coefficient, added together, multiplied by 10 and added to 50.
  Scores on a Scale | 48.2 [36.8 to 81.3]

OUTCOME MEASURES:

1. Primary Outcome: Body Weight Average 6 Months Post-Procedure
Description: The mean body weight of all 5 participants at 6-Months post-procedure.
Time Frame: 6-Month
Measure: Mean (Full Range); unit: lbs.
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
lbs. | 237.6 [161 to 268]

2. Primary Outcome: Body Weight Average 12 Months Post-Procedure
Description: The mean body weight of all 5 participants at 12-Months post-procedure.
Time Frame: 12-Month
Measure: Mean (Full Range); unit: lbs.
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
lbs. | 238 [151 to 272]

3. Primary Outcome: Change in Average Body Weight From Baseline at 6 Months Post-Procedure
Description: Average change in body weight lost.
  Calculated as the average of participants:
  (6-Month Post-Procedure Weight in lbs.) - (Baseline Weight in lbs.)
Time Frame: Baseline, 6 Months
Measure: Mean (Full Range); unit: lbs
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
lbs | 16.6 [2 to 38]

4. Primary Outcome: Change in Average Body Weight From Baseline at 12 Months Post-Procedure
Description: Average change in body weight lost.
  Calculated as the average of participants:
  (12-Month Post-Procedure Weight in lbs.) - (Baseline Weight in lbs.)
Time Frame: Baseline, 12 Months
Measure: Mean (Full Range); unit: lbs
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
lbs | -16.2 [-48 to 0]

5. Primary Outcome: Percentage of Excess Body Weight Loss at 6 Months Post-Procedure
Description: Calculated as the average of participants:
  (((Baseline Weight in lbs.) - (6 Month Post-Procedure Weigh in lbs.))/((Baseline Weight in lbs.) - (Ideal Body Weight in lbs.)))
Time Frame: Baseline, 6 Month
Measure: Mean (Full Range); unit: Percentage of Excess Body Weight Loss
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Percentage of Excess Body Weight Loss | 14.8 [1.8 to 40.4]

6. Primary Outcome: Percentage of Excess Body Weight Loss at 12 Months Post-Procedure
Description: Calculated as the average of participants:
  (((Baseline Weight in lbs.) - (12 Month Post-Procedure Weigh in lbs.))/((Baseline Weight in lbs.) - (Ideal Body Weight in lbs.)))
Time Frame: Baseline, 12 Month
Measure: Mean (Full Range); unit: Percentage of Excess Body Weight Loss
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Percentage of Excess Body Weight Loss | 15.1 [0 to 51.1]

7. Primary Outcome: Average Ghrelin Hormone Levels at 6 Months Post-Procedure
Description: The mean of participant's 6-Month post-procedure Ghrelin levels.
Time Frame: 6-Month
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
pg/mL | 605.4 [331 to 1084]

8. Primary Outcome: Average Ghrelin Hormone Levels at 12 Months Post-Procedure
Description: The mean of participant's 12-Month post-procedure Ghrelin levels.
Time Frame: 12-Month
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
pg/mL | 21.1 [4 to 39]

9. Primary Outcome: Percentage Change in Ghrelin Hormone Levels From Baseline at 6 Months Post-Procedure
Description: Calculated as the average of participants:
  (((6-Month Post-Procedure Ghrelin levels in pg/mL) - (Baseline Ghrelin levels in pg/mL))/(Baseline Ghrelin levels in pg/mL) * 100
Time Frame: 6-Month, Baseline
Measure: Mean (Full Range); unit: Percentage of Change in Ghrelin
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Percentage of Change in Ghrelin | -9.9 [-70.7 to 39.1]

10. Primary Outcome: Percentage Change in Ghrelin Hormone Levels From Baseline at 12 Months Post-Procedure
Description: Calculated as the average of participants:
  (((12-Month Post-Procedure Ghrelin levels in pg/mL) - (Baseline Ghrelin levels in pg/mL))/(Baseline Ghrelin levels in pg/mL) * 100
Time Frame: 12-Month, Baseline
Measure: Mean (Full Range); unit: Percentage of Change in Ghrelin
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Percentage of Change in Ghrelin | -19.2 [-63.6 to 35.9]

11. Secondary Outcome: Average Leptin Hormone Levels at 6 Months Post-Procedure
Description: The mean of participant's 6-month post-procedure Leptin levels.
Time Frame: 6-Month
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
ng/mL | 19.4 [7 to 46.8]

12. Secondary Outcome: Average Leptin Hormone Levels at 12 Months Post-Procedure
Description: The mean of participant's 12-month post-procedure Leptin levels.
Time Frame: 12-Month
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
ng/mL | 21.1 [4 to 39]

13. Secondary Outcome: Percentage Change in Leptin Hormone Levels From Baseline at 6 Months Post-Procedure
Description: Calculated as the average of participants:
  (((6-Month Post-Procedure Leptin levels in ng/mL) - (Baseline Leptin levels in ng/mL))/(Baseline Leptin levels in ng/mL) * 100
Time Frame: 6-Month, Baseline
Measure: Mean (Full Range); unit: Percentage of Change in Leptin
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Percentage of Change in Leptin | -31.2 [-69.2 to 75.3]

14. Secondary Outcome: Percentage Change in Leptin Hormone Levels From Baseline at 12 Months Post-Procedure
Description: Calculated as the average of participants:
  (((12-Month Post-Procedure Leptin levels in ng/mL) - (Baseline Leptin levels in ng/mL))/(Baseline Leptin levels in ng/mL) * 100
Time Frame: 12-Month, Baseline
Measure: Mean (Full Range); unit: Percentage of Change in Leptin
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Percentage of Change in Leptin | 21.1 [4 to 39]

15. Secondary Outcome: Average Cholecystokinin (CCK) Hormone Levels at 6 Months Post-Procedure
Description: The mean of participant's 6-month post-procedure CCK levels.
Time Frame: 6-Month
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
pg/mL | 32.4 [15 to 76]

16. Secondary Outcome: Average Cholecystokinin (CCK) Hormone Levels at 12 Months Post-Procedure
Description: The mean of participant's 12-month post-procedure CCK levels.
Time Frame: 12-Month
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
pg/mL | 44.6 [15 to 73]

17. Secondary Outcome: Percentage Change in Cholecystokinin (CCK) Hormone Levels From Baseline at 6 Months Post-Procedure
Description: Calculated as the average of participants:
  (((6-Month Post-Procedure CCK levels in pg/mL) - (Baseline CCK levels in pg/mL))/(Baseline CCK levels in pg/mL) * 100
Time Frame: 6-Month, Baseline
Measure: Mean (Full Range); unit: Percentage of Change in CCK
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Percentage of Change in CCK | -15.1 [-70.3 to 100]

18. Secondary Outcome: Percentage Change in Cholecystokinin (CCK) Hormone Levels From Baseline at 12 Months Post-Procedure
Description: Calculated as the average of participants:
  (((12-Month Post-Procedure CCK levels in pg/mL) - (Baseline CCK levels in pg/mL))/(Baseline CCK levels in pg/mL) * 100
Time Frame: 12-Month, Baseline
Measure: Mean (Full Range); unit: Percentage of Change in CCK
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Percentage of Change in CCK | 56.4 [-47.0 to 430]

19. Secondary Outcome: Quality of Life (QOL): Averaged Short Form (SF)-36 Version 2 Physical Component Summary (PCS) at 6 Months Post-Procedure
Description: The mean of participant's SF-36 Version 2 PCS at 6 months post-procedure, ranging from 0-100; higher scores indicate better health status. The SF-36v2 contains 8 sections total which are each calculated into individual scale scores. A z-score is then determined for each scale score by subtracting the mean scale score of a sample of the national general population from the scale score of the individual participant being analyzed. Each of the 8 z-scores are then multiplied by the PCS scoring coefficient, added together, multiplied by 10 and added to 50.
Time Frame: 6 Month
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Scores on a Scale | 59.5 [41 to 93.8]

20. Secondary Outcome: Changes in QOL (Measured by SF-36v2 PCS) From Baseline at 6 Months Post-Procedure
Description: The mean of participant's SF-36 Version 2 PCS at 6 months post-procedure, ranging from 0-100; higher scores indicate better health status. The SF-36v2 contains 8 sections total which are each calculated into individual scale scores. A z-score is then determined for each scale score by subtracting the mean scale score of a sample of the national general population from the scale score of the individual participant being analyzed. Each of the 8 z-scores are then multiplied by the PCS scoring coefficient, added together, multiplied by 10 and added to 50.
  Changes in QOL (measured by SF-36v2 PCS) are calculated as the average of participants:
  (6-Month Post-Procedure SF-36v2 PCS) - (Baseline SF-36v2 PCS)
Time Frame: 6 Month, Baseline
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Scores on a Scale | 9.7 [3.2 to 14]

21. Secondary Outcome: QOL: Averaged SF-36v2 PCS at 12 Months Post-Procedure
Description: The mean of participant's 12-month post-procedure Short Form-36 Version 2 Physical Component Scores, ranging from 0-100; higher scores indicate better health status.
Time Frame: 12 Month
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Scores on a Scale | 65.79 [40.2 to 95]

22. Secondary Outcome: Changes in QOL (Measured by SF-36v2 PCS) From Baseline at 12 Months Post-Procedure
Description: The mean of participant's SF-36 Version 2 PCS at 12-months post-procedure, ranging from 0-100; higher scores indicate better health status. The SF-36v2 contains 8 sections total which are each calculated into individual scale scores. A z-score is then determined for each scale score by subtracting the mean scale score of a sample of the national general population from the scale score of the individual participant being analyzed. Each of the 8 z-scores are then multiplied by the PCS scoring coefficient, added together, multiplied by 10 and added to 50.
  Changes in QOL (measured by SF-36v2 PCS) are calculated as the average of participants:
  (12-Month Post-Procedure SF-36v2 PCS) - (Baseline SF-36v2 PCS)
Time Frame: 12 Month, Baseline
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Scores on a Scale | 16.0 [2.4 to 59]

23. Secondary Outcome: QOL: Averaged SF-36v2 MCS at 6 Months Post-Procedure
Description: The mean of participant's SF-36 Version 2 MCS at 6-months post-procedure, ranging from 0-100; higher scores indicate better health status. The SF-36v2 contains 8 sections total which are each calculated into individual scale scores. A z-score is then determined for each scale score by subtracting the mean scale score of a sample of the national general population from the scale score of the individual participant being analyzed. Each of the 8 z-scores are then multiplied by the MCS scoring coefficient, added together, multiplied by 10 and added to 50.
Time Frame: 6 Month
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Scores on a Scale | 57 [41.8 to 88.4]

24. Secondary Outcome: Changes in QOL (Measured by SF-36v2 MCS) From Baseline at 6 Months Post-Procedure
Description: The mean of participant's SF-36 Version 2 MCS at 6 months post-procedure, ranging from 0-100; higher scores indicate better health status. The SF-36v2 contains 8 sections total which are each calculated into individual scale scores. A z-score is then determined for each scale score by subtracting the mean scale score of a sample of the national general population from the scale score of the individual participant being analyzed. Each of the 8 z-scores are then multiplied by the MCS scoring coefficient, added together, multiplied by 10 and added to 50.
  Changes in QOL (measured by SF-36v2 MCS) are calculated as the average of participants:
  (6-Month Post-Procedure SF-36v2 MCS) - (Baseline SF-36v2 MCS)
Time Frame: 6 Month, Baseline
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Scores on a Scale | 8.9 [-1.2 to 20.5]

25. Secondary Outcome: QOL: Averaged SF-36v2 MCS at 12 Months Post-Procedure
Description: The mean of participant's SF-36 Version 2 MCS at 12-months post-procedure, ranging from 0-100; higher scores indicate better health status. The SF-36v2 contains 8 sections total which are each calculated into individual scale scores. A z-score is then determined for each scale score by subtracting the mean scale score of a sample of the national general population from the scale score of the individual participant being analyzed. Each of the 8 z-scores are then multiplied by the MCS scoring coefficient, added together, multiplied by 10 and added to 50.
Time Frame: 12 Month
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Scores on a Scale | 63.1 [36.3 to 88.75]

26. Secondary Outcome: Changes in QOL (Measured by SF-36v2 MCS) From Baseline at 12 Months Post-Procedure
Description: The mean of participant's SF-36 Version 2 MCS at 12-months post-procedure, ranging from 0-100; higher scores indicate better health status. The SF-36v2 contains 8 sections total which are each calculated into individual scale scores. A z-score is then determined for each scale score by subtracting the mean scale score of a sample of the national general population from the scale score of the individual participant being analyzed. Each of the 8 z-scores are then multiplied by the MCS scoring coefficient, added together, multiplied by 10 and added to 50.
  Changes in QOL (measured by SF-36v2 MCS) are calculated as the average of participants:
  (12-Month Post-Procedure SF-36v2 MCS) - (Baseline SF-36v2 MCS)
Time Frame: 12 Month, Baseline
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 5
Scores on a Scale | 14.9 [-6.7 to 48.3]

27. Secondary Outcome: 6-Month Post-Procedure Hemoglobin-A1c (HgA1c) Levels
Description: HgA1c Levels of diabetic patient 6-Months post-procedure.
Time Frame: 6-Month
Population: Applies to the sole diabetic patient in the trial.
Measure: Number; unit: Percentage of HgA1c
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 1
Percentage of HgA1c | 6.3

28. Secondary Outcome: 12-Month Post-Procedure HgA1c Levels
Description: HgA1c Levels of diabetic patient 12-Months post-procedure.
Time Frame: 12-Month
Population: Applies to the sole diabetic patient in the trial.
Measure: Number; unit: Percentage of HgA1c
Arm/Group | Embolic Agent - BeadBlock
Number analyzed (Participants) | 1
Percentage of HgA1c | 5.9

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Embolic Agent - BeadBlock
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Embolic Agent - BeadBlock (N=5)
Mild Nausea, Vomiting (Gastrointestinal disorders) | 2 (2) — Patients 2 and 4 experienced mild nausea, vomiting, mild epigastric discomfort for 24 hours. Superficial gastric ulcers at 3-Day post-procedure endoscopy completely healed at 30-Day post-procedure endoscopy.
Mild Nausea, Vomiting (Gastrointestinal disorders) | 1 (1) — Patient 3 experienced mild nausea, vomiting, mild epigastric discomfort for 3-4 days. Superficial gastric ulcers at 3-Day post-procedure endoscopy completely healed at 30-Day post-procedure endoscopy.

LIMITATIONS AND CAVEATS:
Limitations included:

1. Relatively Small Sample Size
2. Surgical Placebo Effect
3. Lack of Maintaining Diet and Caloric Intake Records
4. Diet Modification and Nutritional Supervision that could account for weight loss

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2014-09-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT02248688/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT02248688/SAP_001.pdf
  • Informed Consent Form (2014-09-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT02248688/ICF_002.pdf